CLINICAL TRIAL: NCT03834597
Title: GlideScope® Versus Macintosh Laryngoscope for Post-thyroidectomy Assessment of Vocal Cord Mobility
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Marwa Ahmed Khairy Elbeialy, Lecturer of Anesthesia, Ain Shams University
Other Study IDs: FMASU R 08/2019
Record Dates: First submitted 2019-02-06; First posted 2019-02-08 (Actual); Last update posted 2019-02-08 (Actual); Status verified 2019-02

CONDITIONS: Complication, Postoperative
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: conventional Macintosh laryngoscope — After closure of surgical, anesthesiologist will perform the conventional Macintosh laryngoscope to assess post-thyroidectomy vocal cord mobility.
Device: GlideScope® — Patient will be left for a while until hemodynamic stabilization then examination with GlideScope® will be commenced to assess postthyroidectomy vocal cord mobility by another experienced anesthesiologist

SUMMARY:
Vocal cord dysfunction is a serious post-thyroidectomy complication. This can lead to various postoperative clinical consequences as hoarseness of voice, aspiration or stridor . It is also one of the common reasons for post-thyroidectomy malpractice claims.

This study will compare GlideScope® with Macintosh laryngoscope regarding accuracy of assessment of post-thyroidectomy vocal cord mobility.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status I and II,
* Elective thyroid surgery with
* Normal thyroid profile

Exclusion Criteria:

* History of previous thyroid surgery,
* Preoperative vocal cord dysfunction
* Predicted difficult airway

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients undergoing elective thyroid surgery
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2019-02-06 (Actual); Primary Completion 2019-05 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Vocal cord dysfunction | Intraoperative
  newly recorded reduction in the postoperative vocal cords mobility compared with the preoperative status.

SECONDARY OUTCOMES:
Incidence of traumatic complications | First 24 hours postoperatively
  traumatic complications as swelling in the mouth, tongue, or throat, teeth injury, bleeding or hoarseness of voice

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided